CLINICAL TRIAL: NCT05706727
Title: Comparative Analytical Study of Intravenous Bolus Dose of Mephentermine and Phenylephrine for Hemodynamic Stability During Elective Cesarean Section Under Spinal Anesthesia at KIST Medical College and Teaching Hospital
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: KIST Medical and Teaching Hospital (Other)
Collaborators: Nepal Health Research Council (Other Government)
Responsible Party: Principal Investigator, Dr. Raju Bikram Basnet, Post Graduate, KIST Medical and Teaching Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: KISTMTH 01
Record Dates: First submitted 2023-01-23; First posted 2023-01-31 (Actual); Last update posted 2024-10-09 (Actual); Status verified 2024-10

CONDITIONS: Hemodynamic Stability
MeSH Terms: interventions — Mephentermine; Phenylephrine

STUDY DESIGN:
Intervention Model Description: Comparative Interventional
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: The patients will be randomly allocated to the two groups of study by sealed envelope method. Group M patients who will receive intravenous bolus dose of mephentermine 6mg and Group P who will receive intravenous bolus dose of phenylephrine 50 mcg The drug preparations phenylephrine 50mcg/ml and mephenterime 6mg/ml will be done and labelled with code numbers by anesthesia assistant for all the patient and it is provided to anesthesiologist for administration who is not involved in the study as they will not be actively involved in the study nor in the patient care. The other anesthesia assistant or intern will be monitoring and recording information on proformas. Therefore investigator and participant of the study were blinded to the study drugs.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Mephentermine ( M group) (Experimental): Group M
  Interventions: Drug: Intravenous bolus dose of Mephentermine and mephentermine
- Phenylephrine ( P group ) (Experimental): Group P
  Interventions: Drug: intravenous bolus dose of phenylephrine 50 mcg

INTERVENTIONS:
Drug: Intravenous bolus dose of Mephentermine and mephentermine — intravenous bolus dose of mephenteramine 6mg
  Other Names: Mephentermine
  Arms: Mephentermine ( M group)
Drug: intravenous bolus dose of phenylephrine 50 mcg — intravenous bolus dose of phenylephrine 50 mcg
  Other Names: Phenylephrine
  Arms: Phenylephrine ( P group )

SUMMARY:
Hemodynamics changes with spinal anesthesia is mainly due to sympathetic block which causes mainly hypotension & bradycardia. Post spinal hypotension usually leads to various adverse maternal and fetal outcomes. Hence, effective prevention and treatment of maternal hypotension is of great clinical significance. Various studies have been done for the prevention of subarachnoid block induced hypotension but the optimal choice of vasopressors for the maintenance of hemodynamic stability during cesarean under spinal anesthesia is still unclear. The ideal vasopressor would be the one which is reliable and easy to use , has rapid onset, short duration of action, easily tritatable, can potentially be used prophylactically and lack any adverse maternal and fetal impact. Thus, aim of study is to compare the hemodynamic stability of mephenterime and phenylephrine during elective cesarean section under spinal anesthesia. The methodology of the study will be prospective, randomized double blinded study where patient meeting inclusion criteria for the study is divided into two groups ( Group M n=21) and ( Group P n= 21) i.e. Group M receives intravenous bolus of mephentermine 6mg and intravenous bolus of 50mcg. Hemodynamics changes in blood pressure and heart rate will monitored and compared among the study groups receiving intravenous boluses of study drugs. Data will be collected in proforma and saved by entering in the MS- EXCEL as well. Data will be analyzed using the statistical package for the social sciences (SPSS) version 27. The categorical data will be analyzed with Chi-square test and numerical variables of hemodynamic parameters between the study groups will be analyzed using student t- test. P-value < 0.05 will be considered statistically significant.

Hence, mephenterime and phenylephrine effectiveness will be studied for hemodynamic stability during cesarean section under spinal anesthesia

DETAILED DESCRIPTION:
Spinal anesthesia is the most common administered neuraxial anesthetic technique for patient undergoing cesarean section due to its rapid and reliable onset and remains preferred choice for cesarean deliveries. The advantage of spinal anesthesia includes no airway manipulation, profound analgesia and anesthesia, minimal maternal and fetal drug exposure stable hemodynamic parameters (based on level of anesthesia), decrease intraoperative blood loss and provide postoperative pain control. Hemodynamics changes is due to sympathetic block which causes reduction in venous return which further reduces the cardiac output and blood pressure by activation of Bezold Jarisch reflex In addition, the vasodilatory effect due to prostaglandins, progesterone relaxin and nitric oxide during pregnancy and loss of intrinsic sympathetic vascular tone further exaggerated fall of blood pressure with prevalence of 50-90% despite of fluid preload and uterine displacement Various preventive measures like fluid preload , left lateral tilt , left uterine displacement and along with vasopressors such as mephentermine , phenylephrine have been tried to prevent hypotension Phenylephrine is currently recommended as 1st line of vasopressor which acts as alpha 1 agonist with negligible beta action increasing blood pressure due to vasoconstriction whereas it causes dose dependent bradycardia and decrease cardiac output Mephentermine non catecholamine nondirectly acts on both adrenergic alpha and beta receptors and indirectly by releasing norepinephrine and epinephrine that increases blood pressure and augments cardiac output whereas tachyphylaxis may occur rapidly.

This study would help to compare the effectiveness of phenylephrine and mephentermine for maintenance of hemodynamic parameters in patient undergoing cesarean section under spinal anesthesia.

ELIGIBILITY:
Inclusion Criteria:

* Patient undergoing elective cesarean section under spinal anesthesia
* Age between 18-48 years
* ASA class II ( all pregnant are categorized as ASA II)

Exclusion Criteria:

* Patient refusal
* Contraindication to spinal anesthesia like coagulation disorder , localized infection , sepsis, raised intracranial pressure etc
* Patchy spinal block , failed spinal block converting to GA
* Hypersensitivity to any drugs
* High Risk Pregnancy ( preeclampsia, eclampsia, preterm, Gestational Diabetes , etc )

Ages: 18 Years to 48 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — All parturient meeting the study inclusion criteria and receiving sub-arachnoid block for undergoing elective cesarean section at KIST MEDICAL COLLEGE AND TEACHING HOSPITAL
Enrollment: 42 (Actual)
Dates: Start 2023-03-23 (Actual); Primary Completion 2024-04-29 (Actual); Study Completion 2024-05-15 (Actual)

PRIMARY OUTCOMES:
To compare the intravenous bolus dose of mephentermine and phenylephrine for hemodynamic stability during elective cesarean section under spinal anesthesia | 6 months
  To measure systolic blood pressure ( SBP) and diastolic blood pressure ( DBP) of the study groups

SECONDARY OUTCOMES:
To measure Mean Arterial Pressure ( MAP ) of study groups | 6 months
  Mean Arterial Pressure will be measured and compared between study groups
To measure heart rate ( HR) of study group | 6 months
  Heart rate will be measured and compared between study groups

CONTACTS AND LOCATIONS:
Overall Officials: Dr. Smriti Koirala, MD, Principal Investigator — KIST Medical College and Teaching Hospital
Locations (1):
- KIST Medical and Teaching Hospital, Lalitpur, Nepal

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Habib AS. A review of the impact of phenylephrine administration on maternal hemodynamics and maternal and neonatal outcomes in women undergoing cesarean delivery under spinal anesthesia. Anesth Analg. 2012 Feb;114(2):377-90. doi: 10.1213/ANE.0b013e3182373a3e. Epub 2011 Nov 21. PMID 22104076
- [Background] Klohr S, Roth R, Hofmann T, Rossaint R, Heesen M. Definitions of hypotension after spinal anaesthesia for caesarean section: literature search and application to parturients. Acta Anaesthesiol Scand. 2010 Sep;54(8):909-21. doi: 10.1111/j.1399-6576.2010.02239.x. Epub 2010 Apr 23. PMID 20455872
- [Background] Corke BC, Datta S, Ostheimer GW, Weiss JB, Alper MH. Spinal anaesthesia for Caesarean section. The influence of hypotension on neonatal outcome. Anaesthesia. 1982 Jun;37(6):658-62. doi: 10.1111/j.1365-2044.1982.tb01278.x. PMID 7091625
- [Background] Ohpasanon P, Chinachoti T, Sriswasdi P, Srichu S. Prospective study of hypotension after spinal anesthesia for cesarean section at Siriraj Hospital: incidence and risk factors, Part 2. J Med Assoc Thai. 2008 May;91(5):675-80. PMID 18672631
- [Background] Campagna JA, Carter C. Clinical relevance of the Bezold-Jarisch reflex. Anesthesiology. 2003 May;98(5):1250-60. doi: 10.1097/00000542-200305000-00030. No abstract available. PMID 12717149
- [Background] Mohta M, Janani SS, Sethi AK, Agarwal D, Tyagi A. Comparison of phenylephrine hydrochloride and mephentermine sulphate for prevention of post spinal hypotension. Anaesthesia. 2010 Dec;65(12):1200-5. doi: 10.1111/j.1365-2044.2010.06559.x. PMID 21182601
- [Background] Mahajan L, Anand LK, Gombar KK. A randomized double-blinded comparison of ephedrine, phenylephrine and mephentermine infusions to maintain blood pressure during spinal anaesthesia for cesarean delivery: The effects on fetal acid-base status and haemodynamic control. J Anaesthesiol Clin Pharmacol. 2009;25(4):427-32.
- [Background] Chandak A V., Bhuyan D, Singam AP, Patil B. Comparison of bolus phenylephrine, ephedrine and mephentermine for maintenance of arterial pressure during spinal anaesthesia in caesarean section. Res J Pharm Technol. 2021;14(3):1349-52.
- [Background] Nag DS, Samaddar DP, Chatterjee A, Kumar H, Dembla A. Vasopressors in obstetric anesthesia: A current perspective. World J Clin Cases. 2015 Jan 16;3(1):58-64. doi: 10.12998/wjcc.v3.i1.58. PMID 25610851